CLINICAL TRIAL: NCT04806308
Title: The Impact of Intraoperative Stretching Microbreaks on Otolaryngologists
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Philip Zapanta, Associate professor, George Washington University
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: ergonomics
Record Dates: First submitted 2021-03-10; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Postural; Strain
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Cross over study so each participant will have 3 control days without intervention and 3 intervention days with stretching exercise.
  Interventions: Behavioral: Otolaryngology stretching micro-breaks (OSMB)
- Control group (No Intervention): Cross over study so each participant will have 3 control days without intervention and 3 intervention days with stretching exercise.

INTERVENTIONS:
Behavioral: Otolaryngology stretching micro-breaks (OSMB) — Standardized microbreak stretch that is designed to perform intraoperatively within the sterile field at medically convenient 20-40 min intervals throughout each procedure.
  Arms: Intervention group

SUMMARY:
There have been numerous survey-based and observational studies reporting a high percentage of otolaryngologists suffering from work-related musculoskeletal symptoms, in which more than half attributed to poor ergonomics in the operating room. Interventions have been implemented in the past to alleviate ergonomic hazards in general surgery such as intra-operative stretch breaks. However, there has not yet been an intervention done to alleviate ergonomic hazards in otolaryngologists. Our study aims to explore the efficacy of implementing intraoperative stretch breaks and assess their effect on otolaryngologists' practices and musculoskeletal pain.

DETAILED DESCRIPTION:
The study subjects will be recruited voluntarily from George Washington University Hospital otolaryngology attending physicians, residents, and fellows, as well as Children's otolaryngology faculties. Pre-survey will be sent prior to the intervention to obtain background information and baseline ergonomic assessment conducted by physical therapy students. Interventions will include intra-operative stretch breaks that will be implemented by surgeons at their convenient time during the surgery. Post-survey will be sent out to obtain the subjects' experiences after each intervention.

Each survey will be sent via email using a secured third-party vendor, RedCap. Results will be retrieved only by the research assistants listed on the institutional review board (IRB). The survey will not ask for any identifying information and will not publish identifying information. The raw data will be analyzed by the PI and research assistant for publication. The study should take less than a year for data collection and analysis.

ELIGIBILITY:
Inclusion Criteria:

* Otolaryngologists
* Currently practicing

Exclusion Criteria:

* Non-otolarynglogists
* Currently not practicing

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-16 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Body part discomfort | Given before each surgery during control days as a baseline
  Body Part Discomfort is a validated survey with 0-5 score on the neck, shoulder R/L, hand R/L, lower/upper back, knee R/L, foot R/L. 0 with no pain to 5 with high pain.
Body part discomfort | Given before each surgery during intervention days
  Body Part Discomfort is a validated survey with 0-5 score on the neck, shoulder R/L, hand R/L, lower/upper back, knee R/L, foot R/L. 0 with no pain to 5 with high pain.
Body part discomfort | Given after each surgery during control days as a baseline
  Body Part Discomfort is a validated survey with 0-5 score on the neck, shoulder R/L, hand R/L, lower/upper back, knee R/L, foot R/L. 0 with no pain to 5 with high pain.
Body part discomfort | Given after each surgery during intervention days
  Body Part Discomfort is a validated survey with 0-5 score on the neck, shoulder R/L, hand R/L, lower/upper back, knee R/L, foot R/L. 0 with no pain to 5 with high pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Park AE, Zahiri HR, Hallbeck MS, Augenstein V, Sutton E, Yu D, Lowndes BR, Bingener J. Intraoperative "Micro Breaks" With Targeted Stretching Enhance Surgeon Physical Function and Mental Focus: A Multicenter Cohort Study. Ann Surg. 2017 Feb;265(2):340-346. doi: 10.1097/SLA.0000000000001665. PMID 28059962
- [Result] Hallbeck MS, Lowndes BR, Bingener J, Abdelrahman AM, Yu D, Bartley A, Park AE. The impact of intraoperative microbreaks with exercises on surgeons: A multi-center cohort study. Appl Ergon. 2017 Apr;60:334-341. doi: 10.1016/j.apergo.2016.12.006. Epub 2016 Dec 29. PMID 28166893

DOCUMENTS (1):
  • Study Protocol (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/08/NCT04806308/Prot_000.pdf